CLINICAL TRIAL: NCT05533970
Title: Ultrasound-guided Modified Fascia Iliaca Compartment Nerve Block for Arthroscopic Knee Surgery： What is the Optimal Dose of Dexmedetomidine?
Brief Title: Ultrasound-guided H-FICB for Arthroscopic Knee Surgery： What is the Optimal Dose of Dexmedetomidine?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K023
Record Dates: First submitted 2022-09-01; First posted 2022-09-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-09

CONDITIONS: Knee Disease; Quality of Recovery
Keywords: modified fascia iliaca compartment block; visual analogue scale(VAS) score

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.375% ropivacaine+0.5ug/kg Dexmedetomidine 30 ml (Experimental): H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine+0.5ug/kg Dexmedetomidine 30 ml
  Interventions: Procedure: ultrasound-guided high fascia iliaca compartment block
- 0.375% ropivacaine+1ug/kg Dexmedetomidine 30 ml (Experimental): H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine+1ug/kg Dexmedetomidine 30 ml
  Interventions: Procedure: ultrasound-guided high fascia iliaca compartment block
- 0.375% ropivacaine+0.25ug/kg Dexmedetomidine 30 ml (Experimental): H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine+0.25ug/kg Dexmedetomidine 30 ml
  Interventions: Procedure: ultrasound-guided high fascia iliaca compartment block

INTERVENTIONS:
Procedure: ultrasound-guided high fascia iliaca compartment block — H-FICB was guided by ultrasound before general anesthesia. The patient was supine. First, the probe is placed transversely above the groin. Then slide the probe up and down to reveal a clear image of the internal oblique and sartorius muscles. There is a bowtie-like iliac fascia space at the junction of these two muscles. After the scanning, the needle was inserted behind the probe with the tip pointed to the ventral side under the guidance of real-time ultrasound; the tip passed through the skin into the iliac fascia space and advanced to the inguinal ligament. After no blood was extracted, 1 ~ 2 ml of normal saline was firstly injected to determine whether the tip position was correct.

SUMMARY:
Total knee replacement (TKR) is among the most commonly performed orthopedic procedures, and a six-fold increase in the number of TKR cases world-wide is projected within a decade as the aging of the populations . As the number of the TKR procedures increases, various approaches increasing the satisfaction and comfort of the patient and the surgeon are of interest in order to provide improved pain management, in-hospital stay, and recovery with the development of modern anesthesiology and pain management techniques.This study aimed to investigate the clinical effect of ultrasound-guided high fascia iliaca compartment block(H-FICB) in patients undergoing knee arthroscopy and to compare it with the normal method which is femoral nerve block combined with a sciatic nerve block to choose the better way. A double-blind, randomized controlled trial was conducted with 44 patients, aged 18-65 years, ASA I-III, who were scheduled to undergo arthroscopic knee surgery in our hospital were selected, the patients were divided into Group A and Group B by random number table method, with 22 patients in each group. Group A was subjected to the H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine+0.5ug/kg Dexmedetomidine 30 ml. Group B was subjected to the H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine+1ug/kg Dexmedetomidine 30 ml.

The mini-mental State Examination was used to assess all the patients' primary cognitive status one day before surgery. The initial acting time and the degrees of sensory block and motor block were recorded after the nerve block was completed. Perioperative variables were recorded to be compared. The investigators used the visual analog scale to assess patients' pain degree with postoperative, recorded the occurrence of adverse events such as postoperative nausea and vomiting(PONV), delayed emergence from anesthesia, and respiratory depression. The confusion assessment method was used to assess whether patients experienced delirium.

DETAILED DESCRIPTION:
1. Study design and setting 44 patients undergoing arthroscopic knee surgery under general anesthesia, gender, aged 18-65 years, American Society of Anesthesiologists (ASA) physical status I-III. Exclusion criteria: communication and dysfunction (e.g., vision, hearing), cerebrovascular history, local anesthetic allergy, opioid allergy, puncture site infection, abnormal clotting.
2. Subjects Patients were allocated randomly to A group (the Modified Fascia Iliaca Compartment block+0.5ug/kg Dexmedetomidine ) and B group (tthe Modified Fascia Iliaca Compartment block+1ug/kg Dexmedetomidine) according to a computer-generated random number table. All patients and an investigator who was responsible for follow-up during 48 postoperative hours were blinded to the randomization groups. In addition, during preoperative visits, the investigators instructed patients on how to use the patient-controlled intravenous analgesia (PCA) device for pain management, as well as how to use the visual analog scale to evaluate pain at rest and while coughing. All the bispectral index (BIS) value in the present study was maintained between 40 and 60 during surgery. All patients voluntarily signed informed consent.
3. General anesthesia Patients were monitored by electrocardiogram, pulse oximetry, and non-invasive blood pressure (one measurement every 3 min) while entering the operation room. A radial artery catheter was also placed for invasive arterial pressure and blood gas monitoring. The induction of general anesthesia was performed intravenously with sufentanil 0.5 µg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Endotracheal intubation was performed with a double-lumen tube. Sevoflurane was used at a minimal alveolar concentration (MAC) of 0.8-1, remifentanil and propofol were used for the maintenance. Fluid management was at the discretion of the attending anaesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years male and female Scheduled for elective arthroscopic knee surgery The patients volunteered to participate in the study and signed the informed consent

Exclusion Criteria:

* Preexisting neuropathy Coagulopathy Local skin infection Hepatic, renal, or cardiorespiratory failure Local anesthetic allergy Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline visual analogue scale | 30 minutes after extubation and 6 hours and 12 hours
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100. A higher score indicates greater pain intensity. Based on the distribution of pain Visual Analogue Scale scores in post-surgical patients knee replacement, who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Numerical Rating Scale have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
cumulative 24-hour postoperative opioid consumption | 24 hours after surgery
  cumulative 24-hour postoperative opioid consumption

SECONDARY OUTCOMES:
The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale | three month after the operation
  During the patients' visits to the pain clinic in the third and sixth months after surgery, an untrained physician unknowingly assessed them. The assessment included evaluating pain intensity, nature, duration, aggravating and mitigating factors, and analgesic medication. The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale was used as the assessment tool to evaluate chronic neuropathic pain in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Principal Investigator — Ethics Committee of Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No